CLINICAL TRIAL: NCT06308614
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Proof-of-Concept Study to Evaluate the Efficacy and Safety of Estetrol in Postmenopausal Subjects With Female Sexual Arousal Disorder
Brief Title: Estetrol for the Treatment of Female Sexual Arousal Disorder in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Estetra (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIT-Do001-C206
Record Dates: First submitted 2024-01-23; First posted 2024-03-13 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Sexual Dysfunction, Physiological
Keywords: Female Sexual Arousal Disorder; FSAD
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Estetrol (Experimental): 20 mg estetrol monohydrate
  Interventions: Drug: 20 mg estetrol monohydrate
- Placebo (Placebo Comparator): Matching Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 20 mg estetrol monohydrate — Active treatment
  Other Names: E4
  Arms: Estetrol
Other: Placebo — Matching Placebo to E4
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is investigating estetrol (E4) in women after menopause, suffering from sexual arousal disorder. The main question it aims to answer is: is 20 mg estetrol monohydrate effective in the treatment of sexual arousal disorder in women after their menopause. Participants will visit the clinic 7 times and complete a daily diary while receiving estetrol or placebo for 12 weeks. Placebo is a pill that looks the same as estetrol but has no active ingredient. Researchers will compare estetrol and placebo to see if estetrol has an effect on the sexual arousal of the participants.

ELIGIBILITY:
Main Inclusion Criteria:

- Hysterectomized postmenopausal women, ≥40 up to ≤65 years, diagnosed with Female Sexual Arousal Disorder

Main Exclusion Criteria:

* Not willing to stop any hormonal products during their participation in the study
* History of unresolved sexual trauma or abuse that is contributing to any sexual dysfunction problem
* Have experienced a recent major life stress or relationship discord that could interfere with sexual activity
* Clinically significant abnormal gynecological findings
* History of malignancy, with the exception of basal cell or squamous cell carcinoma of the skin
* Systolic BP higher than 140 mmHg, diastolic BP higher than 90 mmHg
* Is judged by the investigator to be unsuitable for any reason

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females, born as females
Enrollment: 82 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2025-03-14 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in feeling concerned by difficulties with sexual arousal, assessed by FSDS-DAO Item 14. | 12 weeks
  FSAD = Female Sexual Arousal Disorder
Change from Baseline to Week 12 in the Sexual Function Questionnaire 28 (SFQ-28) Arousal-Sensation Domain (Questions 6 to 9). | 12 weeks
  FSDS-DAO = Female Sexual Distress Scale-Desire/Arousal/Orgasm

SECONDARY OUTCOMES:
Change from Baseline to Week 12 in arousal and lubrication assessed by Patient Reported Outcomes Measurement Information System (PROMIS) Sexual Function and Satisfaction (SexFS) measures (PROMISSexFS Questionnaire). | 12 weeks
Change from Baseline to Week 12 in sexual function assessed by FSDS-DAO - total score. | 12 weeks
Change from Baseline to Week 12 in sexual function assessed by Percentage of Satisfying Sexual Events (SSE) - captured in arousal electronic diary (ediary). | 12 weeks
Change from Baseline to Week 12 in sexual function assessed by SFQ-28 - total score. | 12 weeks
Change from Baseline to Week 12 in sexual function assessed by PROMIS-SexFS. | 12 weeks
Patient Global Impression of Change (PGIC) at Week 12. | 12 weeks
Change from Baseline to Week 12 in severity of sexual arousal disorder as assessed by Patient Global Impression of Severity (PGIS). | 12 weeks

OTHER OUTCOMES:
Frequency of treatment emergent adverse events (TEAEs) (including treatment-emergent serious adverse events [TESAEs]). | 12 weeks
Blood pressure (systolic and diastolic) at each measured time point. | 12 weeks
Respiratory rate at each measured time point. | 12 weeks
Heart rate at each measured time point. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Estetra Study Site, Mesa, Arizona
  - Estetra Study Site, Phoenix, Arizona
  - Estetra Study Site, Tucson, Arizona
  - Estetra Study Site, Pomona, California
  - Estetra Study Site, San Diego, California
  - Estetra Study Site, Jacksonville, Florida
  - Estetra Study Site, Miami, Florida
  - Estetra Study Site, New Port Richey, Florida
  - Estetra Study Site, Ocoee, Florida
  - Estetra Study Site, Orlando, Florida
  - Estetra Study Site, West Palm Beach, Florida
  - Estetra Study Site, Atlanta, Georgia
  - Estetra Study Site, Chicago, Illinois
  - Estetra Study Site, Omaha, Nebraska
  - Estetra Study Site, Las Vegas, Nevada
  - Estetra Study Site, Albuquerque, New Mexico
  - Estetra Study Site, Cleveland, Ohio
  - Estetra Study Site, Englewood, Ohio
  - Estetra Study Site, Memphis, Tennessee
  - Estetra Study Site, Houston, Texas
  - Estetra Study Site, Salt Lake City, Utah
  - Estetra Study Site, Virginia Beach, Virginia
  - Estetra Study Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided